CLINICAL TRIAL: NCT00625027
Title: The Effect of Telehealth Ontario on Non-urgent Emergency Department Use at The Hospital for Sick Children
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dennis Scolnik, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000004841
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Emergency Department Visit
Keywords: Emergency Department Visit; Telehealth Ontario; Triage Levels
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Children presenting to the Emergency Department under the care of a parent or guardian, between 0600 and 2400 during the study period.
  Interventions: Other: Survey and Chart Review

INTERVENTIONS:
Other: Survey and Chart Review — After obtaining consent the survey will be completed. After a staff physician has assessed the patient, the chart will be consulted to retrieve the triage notes, diagnosis, treatment, and discharge recommendations. The physician will be asked to comment on the 'urgency' of the complaint and whether the patient would have been treated equally well at a walk-in clinic.

SUMMARY:
The purpose of this study is to compare the rate of non-urgent emergency department use between three groups of patients: those who were referred to the emergency department by Telehealth Ontario; those who were referred by a physician; and those who arrived without being advised by a nurse or a doctor.

DETAILED DESCRIPTION:
Some studies have shown that certain telephone nursing advice lines are effective in reducing non-urgent emergency department use. However, to my knowledge, no study has investigated the efficacy of Telehealth Ontario in particular. There are important differences between Telehealth Ontario and other phone lines that have been evaluated, in terms of the method in which calls are handled, the diversity of the population served, and the place of the phone-in line within the health care system. These studies, the results of which cannot be extrapolated directly to Telehealth Ontario, should not replace the direct study of the impact and utility of Telehealth Ontario.

Currently Telehealth Ontario receives over 3000 calls daily from residents of Ontario who are concerned about their health. These callers rely on the advise of Telehealth nurses to direct the care they seek out for themselves and for their families. The provincial government also relies on Telehealth Ontario - to provide a useful service within the health care system, relieving the pressure on over-crowded emergency departments by directing patients with non-urgent medical complaints to more appropriate avenues of treatment. This will be the first study to examine the impact of Telehealth Ontario. Although only a small aspect of Telehealth's impact will be examined - the impact on non-urgent emergency department use at Sick Kids - it is an important first step. The results of this study may serve to guide modifications to Telehealth that will make it more accessible to specific groups within the community, more reliable in the advice it provides, and more effective in delivering its message to callers.

ELIGIBILITY:
Inclusion Criteria:

All children presenting to the ED between 0600 and 2400 during the study period

Exclusion Criteria:

1. Children arriving without an adult, as consent could not be obtained.
2. Children with whose parents communication was not possible in English, as it was not possible to provide translation services for this study.
3. Children arriving by direct transfer from another hospital.
4. Children arriving by ambulance summoned by someone other than the parent or guardian.
5. Children arriving at the ED for a pre-arranged visit/appointment.
6. Children requiring immediate resuscitation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children presenting to the ED between 0600 and 2400 during the study period
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The triage categories among patients who did or did not have contact with a health care professional prior to arrival in the ED. | At time of visit to the ED

SECONDARY OUTCOMES:
The demographic and other details of patients arriving with urgent compared to non- urgent complaints. | At time of visit to the ED

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Scolnik, MB ChB, Study Chair — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada